CLINICAL TRIAL: NCT07209124
Title: Increasing Engagement and Positive Emotional Behavior of Older Adults With Mild-Moderate Dementia With the Use of Motion-Based Technology and Meaningful Activities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Collaborators: Community Adult Day Center (Unknown)
Responsible Party: Principal Investigator, Lisa Knecht-Sabres, Professor, Occupational Therapy Program, Midwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB 24028
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Dementia
Keywords: Occupational Therapy; Dementia; Adult Day Care; Engagement; Motion-Based Activities
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The researchers propose to use a randomized control study with a crossover design. More specifically, half of the participants will be randomly assigned to the control group and will engage in the regularly scheduled activities offered at CADC for a 10-week period of time. The other half of the participants will serve as the experimental group and will be randomly allocated to the AB or BA sequence. The participants in the AB sequence will receive treatment A (self-selected Wii games) in the first period (first 5-weeks), and then they will receive treatment B (participation in the Magic Table) in the second period (last 5 weeks). The participants assigned to the BA sequence will participate in treatment B first (Magic Table for the first 5 weeks) and then treatment A (self-selected Wii games) for the last 5 weeks. The researchers will compare scores for all 3 groups on the Assessment of Quality of Activities (A-QOA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention 1 (AB): Engagement in Motion-Based Activities (Wii & Magic Table) (Experimental): The researchers are proposing to use a randomized control study with a crossover design. More specifically, half of the participants will serve as the experimental group and will be randomly allocated to the AB or BA sequence. The participants in the AB sequence will receive treatment A (self-selected Wii games) in the first period (first 5-weeks), and then they will receive treatment B (participation in the Magic Table) in the second period (last 5 weeks). The participants assigned to the BA sequence will participate in treatment B first (Magic Table for the first 5 weeks) and then treatment A (self-selected Wii games) for the last 5 weeks. The researchers will compare scores for all 3 groups on the Assessment of Quality of Activities (A-QOA), to assess the strength of engagement in an activity.
  Interventions: Other: Experimental: Intervention 1 (AB): Engagement in Motion-Based Activities (Wii & Magic Table)
- Intervention 2 (BA): Engagement in Motion-Based Activities (Magic Table BA) (Experimental): The researchers are proposing to use a randomized control study with a crossover design. More specifically, half of the participants will serve as the experimental group and will be randomly allocated to the AB or BA sequence. The participants in the AB sequence will receive treatment A (self-selected Wii games) in the first period (first 5-weeks), and then they will receive treatment B (participation in the Magic Table) in the second period (last 5 weeks). The participants assigned to the BA sequence will participate in treatment B first (Magic Table for the first 5 weeks) and then treatment A (self-selected Wii games) for the last 5 weeks. The researchers will compare scores for all 3 groups on the Assessment of Quality of Activities (A-QOA), to assess the strength of engagement in an activity.
  Interventions: Other: Experimental: Intervention 2 (BA): Engagement in Motion-Based Activities (Magic Table BA)

INTERVENTIONS:
Other: Experimental: Intervention 1 (AB): Engagement in Motion-Based Activities (Wii & Magic Table) — Group to receive treatment/intervention in the AB schedule - Wii first and then magic table
  Arms: Intervention 1 (AB): Engagement in Motion-Based Activities (Wii & Magic Table)
Other: Experimental: Intervention 2 (BA): Engagement in Motion-Based Activities (Magic Table BA) — Group go receive treatment in the BA schedule -- magic table first and then Wii
  Arms: Intervention 2 (BA): Engagement in Motion-Based Activities (Magic Table BA)

SUMMARY:
The purpose of this study is to investigate if engagement in self-selected motion-based games such as Wii and the "Magic Table" is correlated to higher levels of engagement and more positive emotional behaviors.

Individuals may be able to participate in this study if they are an attendee at Community Adult Day Care (CADC) and have a diagnosis of mild-moderate dementia. Individuals need to be able to speak and understand English. Individuals cannot participate if they don't speak English, if they do not attend CADC, or if they have not been diagnosed with mild-moderate dementia Participants will be asked to engage in various activities at the CADC. Participants will be assigned to either the group that will engage in motion-based games such as the Wii gaming system or the Magic Table or will be assigned to a group that engages in typical activities offered by the CADC. If you participate, we will ask you to attend 10 different study-related activity sessions. Each session will last approximately 2 hours and will occur one time per week over approximately 10-weeks.

A potential direct benefit of participating in this study could be that you might have improved mood, behaviors, and/or feelings related to satisfaction and/or quality of life. Involvement in activities also have the potential to improve physical, cognitive, and social skills/function.

The physical risks are minimal and no more than what is expected in routine life and part of everyday activities offered to clients at the CADC.

There is a small chance that involvement in some of the activities may lead to possible feelings of sadness or unease if you are not successful in the desired activity. However, the researchers will do everything possible to modify the activities to enhance success and enjoyment! If any of the activities make you feel uncomfortable, you can stop at any time. You can choose to watch other participants, take a break, or choose not to participate. You do not have to do anything they do not want to do.

If you decide not to participate in this study, you will go about the regularly scheduled programs and activities offered at CADC and no data will be collected for that individual.

DETAILED DESCRIPTION:
This study aims to investigate engagement in self-selected motion-based technology (e.g., Wii and "Magic Table" activities compared to engagement in the everyday activities offered at Community Adult Daycare Center (CADC) correlates with increased engagement and positive behaviors of older adults with mild to moderate dementia. This research will be conducted at CADC in Downers Grove, Illinois. The study will consist of approximately 20 older adults with mild-moderate dementia. The participants will be recruited from CADC on a strictly voluntary basis. Letters of consent and assent will be obtained before the gathering of any data. A letter of support has been obtained from the executive director of CADC. The researchers are proposing to use a randomized control study with a crossover design. More specifically, half of the participants will be randomly assigned to the control group and will engage in the regularly scheduled activities offered at CADC for 10 weeks. The other half of the participants will serve as the experimental group and will be randomly allocated to the AB or BA sequence and will switch after 5 weeks to engage in self-selected activities on both the 'Magic Table' and Wii gaming system. The Assessment of Quality of Activities (A-QOA) observational tool will be filled out weekly by the researchers for each participant to assess their engagement in the activities they are participating in. Higher scores represent more engagement in the activity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals are able to participate in this study if they are an attendee at Community Adult Day Care (CADC) and have a diagnosis of mild-moderate dementia. Participants need to be able to speak and understand English.

Exclusion Criteria:

* Individuals cannot participate if they don't speak English, if they do not attend CADC, or if they have not been diagnosed with mild-moderate dementia.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The Assessment of Quality of Activities (A-QOA) | The Assessment of Quality of Activities (A-QOA) observational tool will be filled out weekly by the researchers over a 10-week period of time for each participant to assess their engagement in the activities they are participating in.
  The Assessment of Quality of Activities (A-QOA) observational tool which assesses engagement in the activities. Higher scores represent more engagement in the activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern University, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogawa M, Shirai H, Nishida S, Tanimukai H. Rasch Analysis of the Assessment of Quality of Activities (A-QOA), an Observational Tool for Clients With Dementia. Am J Occup Ther. 2021 Jan-Feb;75(1):7501205040p1-7501205040p9. doi: 10.5014/ajot.2021.039917. PMID 33399052